CLINICAL TRIAL: NCT04683276
Title: Impact of the Inverted Internal Limiting Membrane Flap Diameter on Idiopathic Macular Hole Closure: Comparative Randomized Study
Brief Title: ILM Inverted Flap Size in Macular Hole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILM flap size
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Idiopathic Macular Hole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- small flap medium-sized macular hole (SFMM) (Active Comparator): small flap (1-2 disc-diameter) was performed in medium sized macular hole (250-400 um)
  Interventions: Procedure: pars plana vitrectomy with ILM inverted flap
- large flap medium-sized macular hole (LFMM) (Active Comparator): large flap (3-4 disc-diameter) was performed in medium sized macular hole (250-400 um)
  Interventions: Procedure: pars plana vitrectomy with ILM inverted flap
- small flap large-sized macular hole (SFLM) (Active Comparator): small flap (1-2 disc-diameter) was performed in Large sized macular hole (>400 um)
  Interventions: Procedure: pars plana vitrectomy with ILM inverted flap
- large flap Large-sized macular hole (LFLM) (Active Comparator): large flap (3-4 disc-diameter) was performed in large sized macular hole (>400 um)
  Interventions: Procedure: pars plana vitrectomy with ILM inverted flap

INTERVENTIONS:
Procedure: pars plana vitrectomy with ILM inverted flap — Complete vitrectomy was done with the aid of triamcinolone acetonide followed by fluid-air exchange. Staining of the ILM was carried with 0.05% solution of Brilliant Blue dye (BBG), (Ocublue plus, Aurolab, India) for 30 seconds, ILM peeling was proceeded leaving a circle of ILM measuring approximately 1-2 DD in SF groups and >2 to 4DD in LF group, centered around the MH. The ILM outside the parafoveal area was peeled to the arcade. The ILM around the hole was then detached from the retina up to the edge of the hole. The ILM flap around the edge of the hole was inverted over the MH using a scraper.

SUMMARY:
In the current study, the investigators described the results of a randomized, comparative clinical trial that was conducted to study the impact of the size of internal limiting membrane (ILM) inverted flap on rate and timing of idiopathic macular hole closure.

DETAILED DESCRIPTION:
A prospective randomized comparative study included patients with idiopathic macular hole (MH) attending outpatient clinic.Eligible eyes were divided into 2 groups based on the narrowest diameter of the MH measured by spectral domain optical coherence tomography (SD-OCT). MHs from 250 to 400µm were classified as Medium-sized MHs and MHs > 400 µm were classified as Large-sized MHs. Within each group, eyes were randomly assigned to either small-flap (1-2DD) or large flap (from >2 to 4DD).

ELIGIBILITY:
Inclusion Criteria:

* Eyes with stage 4 idiopathic MHs with a diameter >250µm on spectral domain optical coherence tomography (SD-OCT)

Exclusion Criteria:

* traumatic MH
* myopic MHs,
* MH secondary to retinal detachment,
* long-standing MH> 12 months
* previous retinal surgeries
* high myopia with an axial length > 26.0 mm
* other ocular pathologies interfering with the interpretation of the OCT reports.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
rate of macular hole closure | 6 months
  defined as the proportion of the eyes with complete MH closure based on SD-OCT findings

SECONDARY OUTCOMES:
timing of MH closure | 6 months
  the time of complete macular hole closure
BCVA | 6 months
  best corrected visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic center, Al Mansurah, Dakahelia, Egypt

IPD SHARING:
Plan to Share IPD: No